CLINICAL TRIAL: NCT06081556
Title: Difference Between Mean Gestational Sac Diameter and Crown-rump Length as a Marker of First-trimester Pregnancy Outcome in Patients With Recurrent Spontaneous Abortion
Acronym: mGSD-CRL& RSA
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: yanlingwork; 81601284 (Other Grant/Funding Number: the National Natural Science Foundation of China)
Record Dates: First submitted 2023-10-07; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Recurrent Spontaneous Abortion
Keywords: recurrent spontaneous abortion; difference between mean gestational sac diameter and crown-rump length; thrombophilia; first-trimester pregnancy outcome
MeSH Terms: conditions — Abortion, Spontaneous; Thrombophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: the difference between mean gestational sac diameter and crown-rump length （mGSD-CRL） ≥ 10mm
  Interventions: Diagnostic Test: ultrasonic testing
- Group B: 10 mm < mGSD-CRL ≤ 15 mm
  Interventions: Diagnostic Test: ultrasonic testing
- Group C: mGSD-CRL >15 mm
  Interventions: Diagnostic Test: ultrasonic testing

INTERVENTIONS:
Diagnostic Test: ultrasonic testing — mean gestational sac diameter（mGSD）, crown-rump length （CRL）, mGSD-CRL, D-dimer (DD), adenosine diphosphate (ADP), arachidonic acid (AA), and the ratio of uterine artery peak systolic value to end-diastolic value (UtA-S/D) were collected
  Other Names: Serum blood test

SUMMARY:
Objective: To determine the effect and predictive value of the difference between the mean gestational diameter (mGSD) sac and crown-rump length (CRL) of the first trimester on the pregnancy outcomes of patients with recurrent spontaneous abortion (RSA).Methods: This is a retrospective cohort study. In total, 256 pregnant women at 6-10 weeks of gestation and with RSA who visited our hospital from January 2020 to March 2023 were included in the study. They were divided into the following three groups based on the difference between the mGSD and CRL (mGSD-CRL): Group A: mGSD-CRL ≥ 10mm, 41 cases; Group B: 10mm < mGSD-CRL ≤ 15mm, 109 cases; and Group C: mGSD-CRL > 15mm, 106 cases.

DETAILED DESCRIPTION:
Study question: Can the difference between mean gestational sac diameter and crown-rump length (mGSD-CRL) act as a marker of first-trimester pregnancy outcome in patients with recurrent spontaneous abortion (RSA)? Summary answer: In patients with RSA, mGSD-CRL acts as an independent risk factor affecting pregnancy outcomes, as it can effectively predict the early pregnancy outcomes of patients with RSA.

What is known already: RSA refers to the occurrence of two or more consecutive miscarriages with the same partner before reaching 28 weeks of gestation, which causes considerable physical and psychological distress to the patients. Therefore, predicting the outcome of subsequent pregnancies in patients with RSA is important. Recent studies have reported a smaller mGSD-CRL difference in association with a higher rate of spontaneous abortion. In addition, thrombophilia-induced RSA has garnered increasing research attention as it is an important cause of early and late miscarriages.

Study design, size, duration: This is a retrospective cohort study. In total, 256 pregnant women at 6-10 weeks of gestation and with RSA who visited our hospital from January 2020 to March 2023 were included in the study. The patients were allocated to three groups based on the mGSD-CRL difference: Group A: mGSD-CRL ≥10 mm, Group B: 10 mm < mGSD-CRL ≤ 15 mm, and Group C: mGSD-CRL >15 mm.

ELIGIBILITY:
Inclusion Criteria:

(1) patients diagnosed with RSA based on medical history, (2) those who intend to continue the pregnancy, (3) singleton pregnancy, (4) gestational age is between 6-10 weeks, and (5) the conception for the current pregnancy was natural

Exclusion Criteria:

(1) individuals with multiple pregnancies or ectopic pregnancies, (2) conception through assisted reproductive techniques, and (3) chromosomal abnormalities in pregnant women or their partners.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — the pregnant women with recurrent spontaneous abortion
Study Population: The pregnant women with RSA who visited the First Affiliated Hospital of Xiamen University from January 2020 to March 2023
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
The pregnancy outcome | The 14 weeks of pregnancy
  The pregnancy outcome at 14 weeks was considered successful if a visible embryo and cardiac activity were confirmed via ultrasound, whereas it was considered a failure if abortion or no cardiac activity was confirmed in the gestational sac by ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Ran, Study Chair — Department of Obstetrics and Gynecology, The First Affiliated Hospital of Xiamen University, School of Medicine, Xiamen University
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
The IPD underlying this article can be made available on reasonable request to the corresponding author.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Yan L, Su Y, Liao Z, Chen H, Ran J. Difference between mean gestational sac diameter and crown rump length predicts pregnancy outcome in patients with recurrent spontaneous abortion. Sci Rep. 2025 Sep 26;15(1):33010. doi: 10.1038/s41598-025-18390-3. PMID 41006676